CLINICAL TRIAL: NCT06332456
Title: Assessment of Renal Microcirculation With Rubidium Positron Emission Tomography: A Proof-of-Concept Study
Brief Title: Assessment of Renal Microcirculation With Rubidium Positron Emission Tomography
Acronym: RESIST
Status: Completed | Type: Observational
Sponsor: Matthieu Pelletier-Galarneau, MD MSc (Other)
Responsible Party: Sponsor-Investigator, Matthieu Pelletier-Galarneau, MD MSc, MD MSc, Montreal Heart Institute
Organization: Montreal Heart Institute (Other)
Other Study IDs: ICM 2023-3169
Record Dates: First submitted 2024-03-14; First posted 2024-03-27 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Renal Microcirculation With Rubidium Positron Emission Tomography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: 15 healthy volunteers
- CKD: 15 patients with CKD and CAD risk factors with GFR between 30 and 45 mL/min/1.73m2

SUMMARY:
The aim of this study is to demonstrate that positron emission tomography imaging with Rubidium-82 (radioactive tracer) can non-invasively detect and quantify changes in renal blood flow (renal perfusion) and renal vascular resistance in both healthy subjects and patients with renal insufficiency. Ultimately, the results of this study will contribute to a better understanding of the role of positron emission imaging in the evaluation of patients with renal diseases.

DETAILED DESCRIPTION:
2. Hypothesis

1. We hypothesize that RBF assessed with rubidium PET is on average lower in patients with CKD. To test our hypothesis, RBF of patients with CKD and coronary artery disease (CAD) risk factors, a population characterized by renal microvascular rarefaction, will be compared to RBF of healthy controls.
2. We hypothesize that RVR assessed with rubidium PET correlates with echographic measurements of renal resistance index (RI), the current non-invasive method of choice.
3. We hypothesize that RBF quantification with rubidium PET is technically reproducible, meaning that the variation on the measurements of RBF purely attributable to technical factors (camera, positioning, tracer injection, etc.) is relatively small. To test this hypothesis, two PET scans will be acquired within a short time period.

3. Objectives and Endpoints 3.1. Primary Objective

1) To compare RBF of patients with CKD and CAD risk factors to healthy controls 3.2. Secondary Objectives

1. To compare RVR of patients with CKD and CAD risk factors to healthy controls
2. To evaluate the correlation between RVR measured with PET to renal RI as measured with echography
3. To evaluate the repeatability and reproducibility of in vivo measurements of RBF and RVR

ELIGIBILITY:
Inclusion Criteria:

Control Group

1. Age ≥ 18 years and < 80 years
2. Signed informed consent
3. No medical history of renal disease

CKD Group

1. Age ≥ 18 years and < 80 years
2. Signed informed consent
3. GFR between 30 and 45 mL/min/1.73m2 measured within the last 3 months
4. At least two cardiovascular disease risk factors such as hypertension, smoking, diabetes, obesity, and dyslipidemia

Exclusion Criteria:

Control Group

1. Hypertension
2. Diabetes
3. Dyslipidemia
4. Active smoking within the last 12 month
5. Left ventricular ejection fraction <45%
6. BMI >45 kg/m2
7. Severe aortic stenosis

CKD Group

1. Left ventricular ejection fraction <45%
2. BMI >45 kg/m2
3. Severe aortic stenosis
4. Changes in medical therapy within the last 4 weeks
5. Documented renal artery stenosis
6. Known structural cause of CKD including polycystic kidney disease, obstruction, or other post-renal causes
7. Pregnancy or breastfeeding
8. Renal failure requiring dialysis within the last 90 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. 15 healthy volunteers
  2. 15 patients with CKD and CAD risk factors with GFR between 30 and 45 mL/min/1.73m2 from HFpEF clinic at ICM
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Renal blood flow in units of mL/min/100g | 1 day
  Average difference of RBF between healthy controls and CKD participants

SECONDARY OUTCOMES:
Renal vascular resistance in units of mmHg/mL/min/100g | 1 day
  Average difference of RVR between healthy controls and CKD participants
Correlation between renal vascular resistance measured with PET and measured with echography | Up to 4 weeks
  Correlation coefficient between RBF vs echographic measurements of renal RI
Coefficient of repeatability of renal blood flow | 1 day
  Coefficient of repeatability, coefficient of variation, and correlation between repeated measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided